CLINICAL TRIAL: NCT06730386
Title: A First-in-human, Phase I Study of Evaluating Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of AK138D1 in the Treatment of Advanced Solid Tumors
Brief Title: A Phase I Study of AK138D1 in the Treatment of Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK138D1-101
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Solid Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK138D1 (Experimental): AK138D1 will be administered in pre-specified dose levels.
  Interventions: Drug: AK138D1

INTERVENTIONS:
Drug: AK138D1 — Enrolled subjects will receive intravenous infusion (IV) of AK138D1 according to the dosing regimen specified in their cohort.

SUMMARY:
This is an open-label, first-in-human, Phase I clinical study aimed at evaluating the safety, tolerability, PK, immunogenicity, and preliminary antitumor efficacy of AK138D1 in subjects being treated for advanced solid tumors.

DETAILED DESCRIPTION:
This study is comprised of two parts: the dose-escalation and dose-expansion stages. Dose-escalation stage aims to determine the MTD/MAD, while the dose-expansion stage is designed to establish the RP2D.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must sign the written informed consent form (ICF) voluntarily;
2. At enrollment, aged ≥ 18 to ≤ 75 years, both males and females are eligible;
3. ECOG performance status score of 0 or 1;
4. Has a life expectancy of ≥ 3 months;
5. Subjects who have histologically or cytologically diagnosed locally advanced or metastatic solid tumor, which Is refractory to or intolerant to standard treatment;
6. At least 1 measurable lesion as per RECIST v1.1 that is suitable for repeated accurate measurement.
7. Adequate organ function.

Exclusion Criteria:

1. Prior human epidermal growth factor receptor 3 (HER3) -targeted therapies, including antibodies, antibody-drug conjugates (ADCs), chimeric antigen receptor T-cell immunotherapy (CAR-T), and others;
2. Concomitant participation in another clinical study, unless it is a non-interventional clinical study or the follow-up period of an interventional study;
3. Presence of active central nervous system (CNS) metastases.
4. Patients with a history of non-infectious pneumonitis requiring systemic corticosteroid therapy; a history of interstitial lung disease (ILD) (including pulmonary fibrosis or radiation pneumonitis); currently suffering from ILD/pneumonitis or suspected of having such diseases based on imaging during screening;
5. Live vaccines or attenuated live vaccines administered within 4 weeks prior to the first dose, or planned to be administered during the study; use of inactivated vaccines is allowed;
6. Untreated subjects with active hepatitis B (HBsAg positive and HBV-DNA exceeding 1000 copies/mL (200 IU/mL) and above the lower limit of detection). For HBsAg-positive subjects, anti-hepatitis B therapy is required during the study; subjects with active hepatitis C (HCV antibody positive and HCV-RNA levels above the lower limit of detection) is also an exclusion;
7. Known active pulmonary tuberculosis (TB); subjects with suspected active TB must undergo appropriate clinical assessment to rule out the presence of active disease;
8. Active syphilis infection;
9. Subjects with known allergy to any component of any study drug; and with a history of known severe hypersensitivity reactions to other monoclonal antibodies;
10. Other reasons for ineligibility as evaluated by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2028-02-26 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
AEs | Up to approximately 2 years
  Incidence and severity of participants with adverse events
Dose-limiting toxicity (DLT) | Up to approximately 2 years
  Occurrence of DLTs and determination fo maximum tolerated dose (MTD)

SECONDARY OUTCOMES:
Cmax and Cmin of AK138D1 | Up to approximately 2 years
  AK138D1 serum drug concentrations in subjects at different time points after administration.
Anti-drug antibodies (ADA) | Up to approximately 2 years
  Number of subjects with detectable anti-drug antibodies (ADA).
Objective Response Rate (ORR) assessed by investigator per RECIST v1.1 | Up to approximately 2 years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) , assessed by investigators based on RECIST v1.1.
Disease Control Rate (DCR) assessed by investigator per RECIST v1.1 | Up to approximately 2 years
  Disease control rate (DCR) assessed according to RECIST v1.1.
Duration of response (DoR) assessed by the investigator per RECIST v1.1 | Up to approximately 2 years
  Duration of response (DoR) assessed according to RECIST v1.1.
Time to response (TTR) assessed by the investigator per RECIST v1.1 | Up to approximately 2 years
  Time to response (TTR) is defined as the time to response based on RECIST v1.1.
Progression Free Survival (PFS) assessed by investigator per RECIST v1.1 | Up to approximately 2 years
  PFS is defined as the time from randomization to the first documented disease progression (per RECIST v1.1 criteria) assessed by investigators or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 2 years
  Overall Survival (OS) is defined as the time from randomization to death due to any cause.

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Blacktown Hospital-Blacktwon Cancer and Haematology Centre, Blacktown, New South Wales
  - Macquarie University, North Ryde, New South Wales
  - ICON Cancer Centre South Brisbane, South Brisbane, Queensland
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria